CLINICAL TRIAL: NCT03787264
Title: A Prospective, Open-label, Multicenter Phase-II Trial to Evaluate the Efficacy and Safety of a Sequential Regimen of Bendamustine Followed by GA101 (obinutuzumab), Acalabrutinib (ACP-196) and ABT-199 (venetoclax) in Patients with Relapsed/refractory CLL (CLL2-BAAG Protocol)
Brief Title: Sequential Regimen of Bendamustin-Debulking Followed by Obinutuzumab, Acalabrutinib and Venetoclax in Patients with Relapsed/refractory CLL
Acronym: CLL2-BAAG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: German CLL Study Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLL2-BAAG
Record Dates: First submitted 2018-12-20; First posted 2018-12-26 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2023-11

CONDITIONS: Chronic Lymphoid Leukemia
MeSH Terms: conditions — Leukemia, B-Cell | interventions — Bendamustine Hydrochloride; obinutuzumab; acalabrutinib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BAAG (Experimental): Debulking: 2 debulking cycles (q 28d) of bendamustine will be administered unless the patient has a contraindication or a debulking is not clinically indicated
  Induction: 6 cycles (q 28d) of Obinutuzumab + Acalabrutinib + Venetoclax
  Maintenance: max. 8 cycles (q 84d) of Obinutuzumab + Acalabrutinib + Venetoclax
  Maintenance treatment will be continued until (whichever occurs first):
  * 12 weeks (approx. 3 months) after confirmation of achievement of a CR/CRi and MRD negativity
  * maintenance cycle 8
  * progression of CLL or start of a subsequent therapy
  * unacceptable toxicity
  Interventions: Drug: Bendamustine; Biological: Obinutuzumab; Biological: Acalabrutinib; Biological: Venetoclax

INTERVENTIONS:
Drug: Bendamustine — Debulking: Cycles 1-2: d1+2 - 70mg/m² i.v.
Biological: Obinutuzumab — Induction: Cycle 1: d1 - 100 mg, d1 (or d2) - 900 mg, d8 + d15 - 1000 mg i.v.; Cycle 2 - 6: 1000 mg, d1 i.v.
  Maintenance: Cycle 1 - 8: 1000 mg, d1 i.v.
  Other Names: GA101; Gazyvaro
Biological: Acalabrutinib — Induction: Cycle 1: --; Cycles 2 - 6: d1-28: 2 x 100mg p.o.
  Maintenance: Cycle 1 - 8: d1-84: 2 x 100mg p.o.
  Other Names: ACP-196; Calquence
Biological: Venetoclax — Induction: Cycles 1 + 2: --; Cycle 3: d1-7: 20mg, d8-14: 50mg, d15-21: 100mg, d22-28: 200mg p.o.; Cycle 4 - 6: d1-28: 400 mg p.o.
  Maintenance: Cycle 1 - 8: d1-84: 400 mg p.o.
  Other Names: ABT-199; Venclyxto

SUMMARY:
CLL2-BAAG is a prospective, open-label, multicenter phase-II trial to evaluate the efficacy and safety of a sequential regimen of debulking with bendamustine followed by induction and maintenance with GA101 (obinutuzumab), acalabrutinib (ACP-196) and venetoclax (ABT-199) in patients with relapsed/refractory CLL.

DETAILED DESCRIPTION:
In the CLL2-BAAG trial will be included a total of 46 patients with relapsed or refractory CLL in need of treatment.This trial will evaluate a debulking with two cycles bendamustine (only for patients with a higher tumor load), followed by an induction and a maintenance treatment with obinutuzumab, acalabrutinib and venetoclax in patients with re-lapsed/refractory CLL. The duration of maintenance treatment is depending on MRD levels. This trial combines one old (chemotherapy) and three novel, synergistic (antibody, BTK-inhibitor and Bcl-2 antagonist) principles of action in order to achieve deep and long lasting remissions with a short duration of treatment. Additionally, this trial has an extensive accompanying scientific program aiming at a better understanding of the kinetics of response and clonal evolution of CLL.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed/refractory CLL in need of treatment according to iwCLL (international workshop on CLL) criteria

   In case of a recent previous treatment, patients must have recovered from acute toxicities and treatment regimen must be stopped within the following time periods before start of the study treatment in the CLL2-BAAG trial:
   * chemotherapy ≥ 28 days
   * antibody treatment ≥ 14 days
   * kinase inhibitors, BCL2-antagonists or immuno-modulatory agents ≥ 3 days
   * corticosteroids may be applied until the start of the BAAG-regimen, these have to be reduced to an equivalent of ≤ 20mg prednisolone per day during treatment Please note: Patients with a progression during previous treatment with venetoclax, ibrutinib or another BTK inhibitor, as well as patients with a known resistance mutation (e.g. BTK-/PLCg2) are excluded from study participation. However, patients who progressed after termination of treatment with venetoclax, ibrutinib, other BTK inhibitors and/or obinutuzumab or who stopped treatment due to in-tolerance to ibrutinib are eligible for participation.
2. Adequate renal function, as indicated by a creatinine clearance ≥30ml/min calculated according to the modified formula of Cockcroft and Gault or directly measured with 24 hr. urine collection
3. Adequate hematologic function as indicated by a neutrophil count ≥ 1.0 x 109/L, a hemoglobin value ≥8.0 g/dL and a platelet count ≥ 25 x 109/L, unless directly attributable to the patient´s CLL (e.g. bone marrow infiltration), in this case, platelet count should be ≥ 10 × 109/L.
4. Adequate liver function as indicated by a total bilirubin ≤2x, AST/ALT ≤2.5x the institutional ULN value, unless directly attributable to the patient's CLL or to Gilbert's Syndrome
5. Negative serological testing for hepatitis B (HBsAg nega-tive and anti-HBc negative, patients positive for anti-HBc may be included if PCR for HBV DNA is negative and HBV-DNA PCR is performed every 4 weeks until one year after last dosage of GA101 (obinutuzumab)), negative testing for hepatitis-C RNA and negative HIV test within 6 weeks prior to registration
6. Age ≥ 18 years
7. ECOG (Eastern Cooperative Oncology Group) performance status 0 - 2, ECOG 3 is only permitted if related to CLL (e.g. due to anemia or severe constitutional symptoms)
8. Life expectancy ≥ 6 months
9. Ability and willingness to provide written informed consent and to adhere to the study visit schedule and other proto-col requirements

Exclusion Criteria:

1. (Suspicion of) transformation of CLL (i.e. Richter's trans-formation, pro-lymphocytic leukemia) or central nervous system (CNS) involvement
2. Progression during previous treatment with venetoclax, ibrutinib or another BTK inhibitor, and/or presence of known mutations associated with resistance to therapy, e.g. Bru-ton´s Tyrosine Kinase and Phospholipase C Gamma 2 (PLCg2)
3. Confirmed progressive multifocal leukoencephalopathy (PML)
4. Malignancies other than CLL currently requiring systemic therapies
5. Uncontrolled infection requiring systemic treatment
6. Any comorbidity or organ system impairment rated with a CIRS (cumulative illness rating scale) score of 4, excluding the eyes/ears/nose/throat/larynx organ system1 or any other life-threatening illness, medical condition or organ system dysfunction that - in the investigator´s opinion - could compromise the patients safety or interfere with the absorption or metabolism of the study drugs (e.g, inability to swallow tablets or impaired resorption in the gastrointestinal tract)
7. Significantly increased risk of bleeding according to the investigator´s evaluation, e.g. due known bleeding diathesis (e.g. von-Willebrandt´s disease or hemophilia), major surgical procedure ≤ 4 weeks or stroke/intracranial hemorrhage ≤ 6 months.
8. Requirement of therapy with strong CYP3A4 inhibitors/inducers or anticoagulant with phenprocoumon (marcumar) or other vitamin K-antagonists
9. Use of investigational agents ≤ 28 days prior to start of study treatment, however, kinase inhibitors, BCL2-antagonists and antibody treatment are allowed in accordance with inclusion criterion number 1 (see above).
10. Known hypersensitivity to obinutuzumab (GA101), venetoclax (ABT-199), acalabrutinib (ACP-196) or any of the excipients Please note: Patients with a known hypersensitivity to bendamustine are allowed to participate but will not receive a debulking with bendamustine
11. Pregnant women and nursing mothers (a negative preg-nancy test is required for all women of childbearing potential within 7 days before start of treatment)
12. Fertile men or women of childbearing potential unless:

    * surgically sterile or ≥ 2 years after the onset of menopause, or
    * willing to use two methods of reliable contraception including one highly effective (Pearl Index <1) and one additional effective (barrier) method during study treatment and for 18 months after end of study treatment.
13. Vaccination with a live vaccine ≤ 28 days prior to registration
14. Legal incapacity
15. Prisoners or subjects who are institutionalized by regula-tory or court order
16. Persons who are in dependence to the sponsor or an investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2021-02-11 (Actual); Study Completion 2023-09-26 (Actual)

PRIMARY OUTCOMES:
Negativity rate of minimal residual disease (MRD) in peripheral blood (PB) measured by 4-color flow cytometry | At final restaging (RE): 12 weeks after the start of the last induction cycle
  MRD negativity is defined as less than one (1) CLL-cell among 10,000 leukocytes analyzed [0.01%], i.e. < 10-4. The MRD negativity rate is defined as the proportion of patients having achieved MRD negativity based on the full analysis set (FAS).

SECONDARY OUTCOMES:
Overall response rate (ORR) | At final restaging (RE): 12 weeks after the start of the last induction cycle
  Proportion of patients having achieved a complete response (CR), a CR with incomplete recovery of the bone marrow (CRi), or a partial response(PR) as best response.
CR / CRi rate | At final restaging (RE): 12 weeks after the start of the last induction cycle
  Proportion of patients having achieved a CR or CRi as best response
MRD in PB measured by 4-color flow cytometry at different times: At screening, after debulking, 4-weekly during induction, at initial response assessment (after 6 induction cycles), at RE, every 12 weeks during maintenance and follow up. | From date of screening until the end of follow-up, up to 40 month.
  MRD negativity is defined as less than one (1) CLL-cell among 10,000 leukocytes analyzed [0.01%], i.e. < 10-4. MRD values will be categorized into negative (<10-4) and positive (≥10-4)
Safety: Adverse events (AE), serious adverse events (SAE) and adverse events of particular interest (AEPI) | up to 40 months after first dose of study drug
  Type, frequency, and severity of AEs, SAEs and AESIs and their relationship to study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Cramer, Dr. med., Principal Investigator — German CLL Study Group
Locations (17):
- Germany (17):
  - Universitätsklinik Köln, Cologne
  - Gemeinschaftspraxis Hämatologie Onkologie, Dresden
  - Gemeinschaftspraxis Mohm/Prange-Krex, Dresden
  - Universitatsklinik Carl Gustav Carus, Dresden
  - Helios Klinikum Erfurt, Erfurt
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Jena, Jena
  - Praxis fuer Haematologie und Onkologie, Koblenz
  - Gemeinschaftspraxis Haemato/ Onkologie Lebach, Lebach
  - Klinikum Leverkusen GmbH, Leverkusen
  - Krankenhaus Muenchen-Schwabing, Munich
  - Ludwig-Maximilians-Universitaet Muenchen, München
  - Praxis Dr. Uhlig, Naunhof
  - Universitätsklinik Rostock, Rostock
  - ZAHO-Rheinland, Siegburg
  - Universitaetsklinik Tuebingen, Tübingen
  - Universitätsklinikum Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Furstenau M, Weiss J, Giza A, Franzen F, Robrecht S, Fink AM, Fischer K, Schneider C, Tausch E, Stilgenbauer S, Ritgen M, Schilhabel A, Bruggemann M, Eichhorst B, Hallek M, Cramer P. Circulating Tumor DNA-Based MRD Assessment in Patients with CLL Treated with Obinutuzumab, Acalabrutinib, and Venetoclax. Clin Cancer Res. 2022 Oct 3;28(19):4203-4211. doi: 10.1158/1078-0432.CCR-22-0433. PMID 35594173
- [Background] Cramer P, Furstenau M, Robrecht S, Giza A, Zhang C, Fink AM, Fischer K, Langerbeins P, Al-Sawaf O, Tausch E, Schneider C, Schetelig J, Dreger P, Bottcher S, Kreuzer KA, Schilhabel A, Ritgen M, Bruggemann M, Kneba M, Stilgenbauer S, Eichhorst B, Hallek M. Obinutuzumab, acalabrutinib, and venetoclax, after an optional debulking with bendamustine in relapsed or refractory chronic lymphocytic leukaemia (CLL2-BAAG): a multicentre, open-label, phase 2 trial. Lancet Haematol. 2022 Oct;9(10):e745-e755. doi: 10.1016/S2352-3026(22)00211-3. Epub 2022 Aug 18. PMID 35988545
- [Background] Furstenau M, Giza A, Weiss J, Kleinert F, Robrecht S, Franzen F, Stumpf J, Langerbeins P, Al-Sawaf O, Simon F, Fink AM, Schneider C, Tausch E, Schetelig J, Dreger P, Bottcher S, Fischer K, Kreuzer KA, Ritgen M, Schilhabel A, Bruggemann M, Stilgenbauer S, Eichhorst B, Hallek M, Cramer P. Acalabrutinib, venetoclax, and obinutuzumab in relapsed/refractory CLL: final efficacy and ctDNA analysis of the CLL2-BAAG trial. Blood. 2024 Jul 18;144(3):272-282. doi: 10.1182/blood.2023022730. PMID 38620072
- See also: Click here for more information about this study: CLL2-BAAG (German CLL Study Group) — https://www.dcllsg.com/cll2-baag/